CLINICAL TRIAL: NCT05201417
Title: Adapted Physical Activity and Prevention of Cardiovascular Risk in Elderly People Living With HIV: Comparative Study of Two Cohortes, CHU Saint Etienne (France) and Mvog Ada District Hospital Yaoundé, Cameroon.
Brief Title: Adapted Physical Activity and Prevention of Cardiovascular Risk in Elderly People Living With HIV:Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Support and Education Technic Centre (Other)
Responsible Party: Principal Investigator, Bienvenu BONGUE, principal investigator, Support and Education Technic Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UJM_UB_01
Record Dates: First submitted 2021-10-31; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Cardiovasculars Risk Factors; Heart Failure
Keywords: adapted physical activity; cardiovascular diseases; Elderly; HIV; Prevention
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group A (No Intervention): patients continue their usual HIV management no intervention
- intervention group B (Other): patients continue their usual HIV management, patients will benefit from an adapted physical activity program for 12 weeks
  Interventions: Other: adapted physical activity

INTERVENTIONS:
Other: adapted physical activity — The adapted physical activity will be administered remotely through the whatsApp or YouTube application. Two sessions will be done per week: Wednesday and Sunday. Walking seems to be appropriate for all participants We will account for 24 APA sessions. We will leverage the Step Tracker phone app and pedometer to get the number of steps done, number of calories spent, Workout duration and distance walked per participant per APA session; this data will be collected weekly (after every two sessions)
  Arms: intervention group B

SUMMARY:
A quasi-experimental and comparative study will be conducted in two different geographical areas (Europe-France and Africa-Cameroon) on a period of 18 months. All eligible adults aged 50 years and older presenting to one of the investigative centers (for HIV care) will be included in the study. The patients will be randomized in two parallel groups according to the 1:1 ratio, namely a control group A where patients continue the usual HIV management, and an intervention group B where in addition to the usual HIV management, patients will benefit from an adapted physical activity (APA) program for three months. An evaluation of heart rate variability, response to current treatment, gut microbiota profile and quality of life will be performed at the end of the APA session. Comparison between control group A and intervention group B will be performed. The acceptability of this program will also be evaluated.

DETAILED DESCRIPTION:
Purpose: The objective of our study was to measure the effect of a physical activity training program on heart rate variability (ANS) in PLWHIV in 2 different geographical areas (Europe-France and Africa-Cameroon). Investigators also propose to measure the impact of this program on inflammation markers such as IL-6, ultra-sensitive CRP and Cystatin C, on the quality of the microbiota of PLHIV and TMAO.

participants and methods: Investigators will conduct a comparative study that involved subjects aged from 50 years and above, recruited from June 2019 to June 2020 at Mvog Ada district hospital

This study will be conducted in 3 phases:

* Phase 1: All eligible adults aged 50 years and older presenting to one of the investigative centers (for HIV care) will be included in the study. The standardized program of adapted physical activity is proposed on the basis of the specifications of adapted physical activities. The participants will be randomized in two parallel groups according to the 1:1 ratio, namely a control group A where participants continue their usual HIV management, and an intervention group B where in addition to the usual HIV management, participants will benefit from an adapted physical activity program. Information regarding heart rate variability and ANS dysfunction will be collected via an overnight recording with the NeuroCoach device (recording box). A questionnaire (to determine the level of physical activity, on compliance with current treatment and quality of life) will be administered.
* Second phase: intervention phase The adapted physical activity program will be offered systematically to all participants in group B. The standardized program of adapted physical activity is proposed on the basis of the specifications of adapted physical activities. An evaluation of heart rate variability, response to current treatment, gut microbiota profile and quality of life will be performed at the end of the APA sessions. Comparison between control group A and intervention group B will be performed.
* The third phase: post-program follow-up: six months At the end of the intervention phase, post-program follow-up will be done through interviews until six months after the end of the intervention. All the participants included will be able to benefit, at their request, a counseling session related to the adapted physical activity program, in order to reinforce integration of physical activity into their day to day routine.

ELIGIBILITY:
Inclusion Criteria:

* People aged 50 to 77 years ;
* People living with HIV in one of the 2 study'countries;
* People without medical contraindications to participate in moderate physical activity
* People who has received information about the study and its rights to its data.

Exclusion Criteria:

* Patient under guardianship or curatorship;
* Having a contraindication to physical activity (medical certificate);
* Infected with HIV-2 alone;
* Hospitalized, in end of life care;
* Morbidly obese (BMI > 40).

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-06-06 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
heart failure | At inclusion and after 24 weeks
  evaluated by summing the participant's factors contributing to heart rate variability. The Neurocoach records a 24-hour electrocardiogram (ECG). From this 24-hour recording, 3 types of variable are given, cardiac arrhythmias, Autonomic nervous system (ANS) activity, Sleep apnea parameters. the punctual analysis of the neurocoach recording makes it possible to highlight atrial fibrillation (AF) and sleep apnea, factors known to promote the risk of a cardiovascular accident
cardiovascular risks factors | At inclusion and after 24 weeks
  evaluated by summing the participant's cardiovascular risk factors. The cardiovascular risk factors assess were metabolic disorders(Total cholesterol, HDL cholesterol, Triglyceride), smoking, physical inactivity, alcohol consumption (defined by an AUDIT score ≥ 8), overweight or obesity, hypertension, and diabetes. The cardiovascular risk was considered high if the subject had a combination of at least 3 cardiovascular risk factors.

SECONDARY OUTCOMES:
total cholesterol ( mg/l) | At inclusion , up to 12 weeks and after 24 weeks
  <190mg/dl = normal and >190 mg/dl = high
HDL cholesterol ( mg/dl) | At inclusion , up to 12 weeks and after 24 weeks
  Men (> 55 mg /dl = normal; 35 - 55 mg/dl = intermidiate; < 35 mg/dl = low ) women (> 65 mg/dl = normal; 45 - 65 mg/dl = intermidiate, < 45 mg/dl = low)
Triglyceride (mg/dl) | At inclusion , up to 12 weeks and after 24 weeks
  Normal: <150 mg/dl, slightly elevated: 150-200mg/dl, high 200 - 500 mg/dl and very high ≥ 500 mg/dl
atrial fibrillation-type heart rhythm disturbances | At inclusion and after 24 weeks
  Atrial fibrillation occurs when action potentials fire very rapidly within the pulmonary veins or atrium in a chaotic manner. Because the atrial rate is so fast, and the action potentials produced are of such low amplitude, P waves will not be seen on the ECG in patients with atrial fibrillation.
  the Neurocoach is worn by the participant overnight, allowing the investigator to analyze their nightly ECG recording.
an indirect approach to the presence of sleep apnea | At inclusion and after 24 weeks
  Heart rate allows to count sleep apnea events. Neurocoach records a 24-hour electrocardiogram (ECG). From this 24-hour recording a sleep apnea are notice throw heart rate decreases due to the stretching of mechanical receptors of the lungs. Once the ventilation resumes, heart rate increases due to the hypoxia stimuli accumulated during the apnea. These swings in heart rate allow to quantify sleep apnea.
  AHI (Apnea/Hypopnea Index): number of breaths stopped (apneas) or number of shallow breaths (hypopneas) per hour of sleep.
  * From 5 to 15 ...... Mild Sleep Apnoea Syndrome
  * 15 to 30 .... Moderate Sleep Apnoea Syndrome
  * More than 30 ..... Severe Sleep Apnoea Syndrome.
disturbances in the activity of the autonomic nervous system | At inclusion and after 24 weeks
  Neurocoach records a 24-hour electrocardiogram (ECG). From this 24-hour recording the variations of the RR intervals which are dependent on the innervation by the Autonomic Nervous System (ANS) which modify the RR intervals on short terms, from one interval to the other, as well as on longer terms.From the analysis of the variations of this intervals, one can deduce the activity of the ANS
  The parasympathetic and sympathetic variables are better separated using Fourier Transform:
  * High Frequency (HF 0,15 et 0,4 Hz.) gives the parasympathetic activity
  * Low frequency (LF 0,04 et 0,15 Hz) gives the sympathetic activity
  * The LF/HF ratio gives the equilibrium between both activities Ratio < 2 .......... balanced sympathetic-vagal balance
  * 2 < Ratio < 4 .... slightly unbalanced sympathetic-vagal balance
  * 4 < Ratio < 6 .... unbalanced sympathetic-vaginal balance
  * 6 < Ratio .......... strongly unbalanced sympathetic-vagal balance
inflammatry marker(Il-6) | At inclusion , up to 12 weeks and after 24 weeks
  nomal range 5-15 pg/ml
Cystatin C (mg/l) | At inclusion , up to 12 weeks and after 24 weeks
  Normal : 0.48 - 0.82 (woman < 60 years) 0.54 - 0.94 (man < 60 years) and 0.63 - 1.03 (≥ 60 years)
ultra sensitive CRP. | At inclusion , up to 12 weeks and after 24 weeks
  Low risk of developing cardiovascular disease (<1.0 mg / l); Average risk of developing cardiovascular disease (1.0 to 3.0 mg / L); High risk of developing cardiovascular disease (3.0-10.0 mg / L); Other cause of inflammation (> 10.0 mg / L)
gut microbiota | At inclusion and after 24 weeks
  Quantification of the most important probiotics in the gut microbiota (Faecalibacterium and Eubacterium) by RT-q PCR
adapted physical activity | 12 weeks
  The adapted physical activity will be administered remotely through the whatsApp or YouTube application. Two sessions will be done per week: Wednesday and Sunday. Walking seems to be appropriate for all participants. We will account for 24 APA sessions. We will leverage the Step Tracker phone application to get the number of steps doneand Workout duration (minute) per APA session; this data will be collected weekly

OTHER OUTCOMES:
Smoking | At inclusion
  answering "yes" to the question do you smoke?
Alcoholism | At inclusion
  answering "yes" to the question do you consume alcohol?
Body mass index | At inclusion
  3 modalities was defined according to BMI. Underweight (BMI < 18.5 Kg/m2), normal weight (18 ≤ BMI < 25 Kg/m²), overweight (25 ≤ BMI < 30 Kg/m²), obesity (BMI ≥ 30 Kg/m²).
Systolic Blood Pressure (mmHg) | At inclusion
  Systolic blood pressure ≥ 140 mmHg or taking a hypotensive treatment.
Diastolic Blood Pressure (mmHg) | At inclusion
  diastolic ≥ 90 mmHg or taking a hypotensive treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ROCHE, professor, Study Chair — 5. University Jean Monnet, St Etienne, Laboratory SNA-EPIS EA 4607, France
Locations (3):
- Mvog Ada district Hospital, Yaoundé, Centre Region, Cameroon
- France (2):
  - CHU Saint-Etienne, Saint-Etienne
  - CHU Saint étienne, Saint-Etienne